CLINICAL TRIAL: NCT03227666
Title: The Effect of Progressive Balance Exercise on Postural Sway - a 4 Week Randomized Controlled Trial
Brief Title: Improving Balance Through Balance Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Västerbotten (Other Government)
Collaborators: Swedish Research Council, Kamprad Family Foundation, Kempe Foundation (Unknown)
Responsible Party: Principal Investigator, Anna Nordström, Adjunct Professor, Region Västerbotten
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: VCC-LIFE-2
Record Dates: First submitted 2017-07-13; First posted 2017-07-24 (Actual); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Balance; Distorted; Fall
Keywords: Postural sway; Progressive balance exercise; RCT; Functional balance
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Intervention group recieving exercise and control group recieving no exercise
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention group will perform three supervised group training sessions a week, consisting of 30 minutes of balance training for 4 weeks.
  Interventions: Behavioral: Exercise
- Control group (No Intervention): The control group recieves a health consultation that highlights the importance of physical activity and balance exercise according to standard practice within the HAI project. They are asked to return after 4 weeks for follow up.

INTERVENTIONS:
Behavioral: Exercise — The intervention group will perform three supervised group training sessions a week, consisting of 30 minutes of balance training for 4 weeks.
  Arms: Intervention Group

SUMMARY:
Today most fracture prevention measures targets the bone and osteoporosis. However, only about 20% of individuals with fractures have osteoporosis and at least 90% of all fractures are caused by a fall. Therefore, the present project builds on previous findings from our group identifying postural sway as an important risk factor for falls and aims to intervene against this risk factor in a randomized controlled trial targeting subjects at the highest risk for falls.

DETAILED DESCRIPTION:
Specific aims:

1. Examine whether four weeks progressive balance training can improve parameters of body sway in measurements of static standing balance
2. Investigate whether participants experience greater security to their own ability and less fear of future falls after 4 weeks of progressive balance training
3. Investigate how long a potential effect of progressive balance training may be noticeable on participants' experiences of greater security in their own ability and less fear of future falls
4. 3. Examine whether participation in balance training leads to reduced number of falls at follow-up after 6, 12 and 24 months

Falls and fall-related injuries are major health concerns for elderly individuals; they cause functional decline and increased mortality, as well as incurring vast health care costs for society. Occurrences and consequences of falls are expected to increase globally with the growing number of elderly individuals. Hence, the improved detection and prediction of potential fall risk markers are of individual and societal importance.

Falling can be the end result of intrinsic and extrinsic factors negatively affecting an individual's ability to maintain balance, which are often revealed during sequences of body movement. Balance can be both dynamically and statically measured, the latter involves having the individual in a stationary standing position, from which results researchers have proposed impaired postural stability as a risk factor for falling. However, evidence regarding the association of postural instability with prospective falls is limited, and population-based cohort studies in this field are scarce. Other shortcomings of previous studies include the use of retrospective study designs, which increase the risks of recall bias and the identification of risk factors as the result of falls.

Postural instability is preferably investigated using objective measures of posturography, the advantages of which over regular clinical assessments include the reduction of test performance variability and avoidance of subjective scoring systems. Recently, researchers have analyzed the performance of the Wii Balance Board (WBB; Nintendo, Kyoto, Japan) in the measurement of postural instability; WBB-based assessment has shown excellent concurrent validity and the ability to complement existing fall assessments.

As of 2012, all 70-year olds in the Umeå municipality are invited to participate in the Healthy Ageing Initiative (HAI) study, which has currently enrolled more than 3000 participants. Among other measurements, we include assessment of postural stability using a Wii Balance Board (WBB; Nintendo, Kyoto, Japan) device. With each participant in a quiet stance, balance trials consisting of 60-second eyes-open (EO) and eyes-closed (EC) trials are performed. Participants are instructed to maintain an upright position throughout the test, stand relaxed, and avoid any arm or head movement. The WBB measures total COP sway length, representing the sum of postural sway in the anteroposterior and mediolateral directions.

Preliminary results from analyses of data consisting of 1900 70-year-old individuals revealed that participants with postural sway in the 5th quintile had almost twice the risk of falling compared to the reference group, when the 1-year follow-up of prospective falls was performed.

Thus the aim of the present follow-up study is to investigate if the investigators can reduce the increased postural sway of participants who have been identified as having abnormal balance values, based on previous measurements.

The present project is planned to be conducted as a 4-week randomized intervention study with a follow up time of 2 years.

Recruitment of participants at high risk of falls from the Healthy Ageing Initiative will be performed. The Healthy Ageing Initiative (HAI) is an ongoing population based project aiming to reduce risk factors for non-communicable diseases (NCD) by risk factor evaluation and increased physical activity. In short, HAI is inviting all 70 year olds in Umeå municipality to a health examination where traditional and potential novel risk factors for diabetes, CVD and fractures are investigated. These include objective measures of physical activity, blood pressure, blood-glucose, objective measured abdominal fat mass and ectopic fat, bone density and other features of bone quality, cognitive function, balance, walking ability, and different life style factors. At the second visit, all participants are informed about the results of tests performed and gets advice with a focus on physical activity, aiming at decreasing the risk of future diabetes, CVD and fractures. The counseling with focus on physical activity is based on motivational interviewing (MI) which is a directive patient-cantered counseling style to help the participants to explore and resolve their ambivalence about behavior change. They are contacted at 6,12 and 24 months per telephone for follow up and are contacted for an in-clinic follow up after 5 years.

Participants in HAI identified as being in the highest quartile of measures of postural sway, indicating poor balance and high fall risk, are invited to participate by telephone contact, and will upon agreement be randomized into either the intervention group or control group. Participants will after the initial contact also receive written information about the study. The investigators aim to recruit 200 individuals from the existing HAI study cohort

After 4 weeks, the participants are followed up with the same measures that are used in the HAI that contains objective and functional balance tests, tests of muscle strength and a validated questionnaires on fear-of-falling and physical activity. Both groups will be offered the specific program for balance training post measurements, with instructions that it can be performed in the home setting according to the same principles offered to the intervention group. The groups are followed up after 6 and 12 months through 70-years-health checks on prospective falls and levels of physical activity.

Descriptive data will be presented as M+SDs and the Student's t-test will be used to analyze statistical differences between variables. Categorical variables are investigated using chi-squared tests. Potential differences between intervention and control group will be analyzed using paired t-tests and two-way repeated measures ANOVA. All analyses will be performed with SPSS version 24 (IBM Corp, Armonk, NY, USA) and Stata version 13.1 (StataCorp, College Station, Texas, USA).

This study could potentially lead to increased understanding of how balance exercise can contribute to an improved balance in individuals with impaired balance and ability. The investigators also intend to highlight the participant's confidence in, and experience of, their own balance ability, and if the fear of future falls is reduced. This is important knowledge in order to prevent falls and fall injuries in older individuals, which are expected to increase in number in society. Through improvements in balance, future falls can potentially be preventable, which contributes to less fall-related injuries and accidents, thereby maintaining functional ability in especially older individuals. The prevention of falls and fall injuries reduces the suffering of individuals, but can also reduce health care costs when care for fall injuries such as hip fractures can be reduced.

ELIGIBILITY:
Inclusion Criteria:

* Participation in the HAI study, having postural sway > 400 mm during Eyes Open trial or > 920 mm during Eyes Closed trial

Exclusion Criteria:

* Walking aid

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-08-12 (Actual); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
Change in Postural Sway | Change in Baseline Postural Sway at 4 weeks
  Total postural sway length, measured objectively during trials of eyes open and eyes closed, during 60 seconds each

SECONDARY OUTCOMES:
Prospective Falls | 6,12 and 24 months after intervention
  Self-recalled during telephone follow-up
Change in Time-up-and-go (TUG) Performance | Change in Baseline TUG Performance at 4 weeks
  Clinical balance test assessing ability to rise from chair, walk back and forth 3 meters and sit back down
Change in Balance Self-efficacy | Change in Baseline Balance Self-efficacy at 4 weeks
  Falls Efficacy Scale (FES)
Change in Fear of Falling (FOF) | Change in Baseline FOF at 4 weeks
  Falls Efficacy Scale International (FES-I)
Change in Muscle Strength | Change in Baseline Muscle Strength at 4 weeks
  Grip strength measured by isokinetic hand dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Anna Nordström, PhD, Principal Investigator — Västerbotten County Council, Umeå University
Locations (1):
- Livsmedicin (LIFE), Umeå, Västerbotten County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stel VS, Smit JH, Pluijm SM, Lips P. Consequences of falling in older men and women and risk factors for health service use and functional decline. Age Ageing. 2004 Jan;33(1):58-65. doi: 10.1093/ageing/afh028. PMID 14695865
- [Background] Wolinsky FD, Fitzgerald JF, Stump TE. The effect of hip fracture on mortality, hospitalization, and functional status: a prospective study. Am J Public Health. 1997 Mar;87(3):398-403. doi: 10.2105/ajph.87.3.398. PMID 9096540
- [Background] Rizzo JA, Friedkin R, Williams CS, Nabors J, Acampora D, Tinetti ME. Health care utilization and costs in a Medicare population by fall status. Med Care. 1998 Aug;36(8):1174-88. doi: 10.1097/00005650-199808000-00006. PMID 9708590
- [Background] Masud T, Morris RO. Epidemiology of falls. Age Ageing. 2001 Nov;30 Suppl 4:3-7. doi: 10.1093/ageing/30.suppl_4.3. No abstract available. PMID 11769786
- [Background] Robinovitch SN, Feldman F, Yang Y, Schonnop R, Leung PM, Sarraf T, Sims-Gould J, Loughin M. Video capture of the circumstances of falls in elderly people residing in long-term care: an observational study. Lancet. 2013 Jan 5;381(9860):47-54. doi: 10.1016/S0140-6736(12)61263-X. Epub 2012 Oct 17. PMID 23083889
- [Background] Tinetti ME, Speechley M, Ginter SF. Risk factors for falls among elderly persons living in the community. N Engl J Med. 1988 Dec 29;319(26):1701-7. doi: 10.1056/NEJM198812293192604. PMID 3205267
- [Background] Maki BE, Holliday PJ, Topper AK. A prospective study of postural balance and risk of falling in an ambulatory and independent elderly population. J Gerontol. 1994 Mar;49(2):M72-84. doi: 10.1093/geronj/49.2.m72. PMID 8126355
- [Background] Piirtola M, Era P. Force platform measurements as predictors of falls among older people - a review. Gerontology. 2006;52(1):1-16. doi: 10.1159/000089820. PMID 16439819
- [Background] Lord SR, Sambrook PN, Gilbert C, Kelly PJ, Nguyen T, Webster IW, Eisman JA. Postural stability, falls and fractures in the elderly: results from the Dubbo Osteoporosis Epidemiology Study. Med J Aust. 1994 Jun 6;160(11):684-5, 688-91. PMID 8202002
- [Background] Moe-Nilssen R, Nordin E, Lundin-Olsson L; Work Package 3 of European Community Research Network Prevention of Falls Network Europe. Criteria for evaluation of measurement properties of clinical balance measures for use in fall prevention studies. J Eval Clin Pract. 2008 Apr;14(2):236-40. doi: 10.1111/j.1365-2753.2007.00839.x. PMID 18324932
- [Background] Howcroft J, Kofman J, Lemaire ED. Review of fall risk assessment in geriatric populations using inertial sensors. J Neuroeng Rehabil. 2013 Aug 8;10(1):91. doi: 10.1186/1743-0003-10-91. PMID 23927446
- [Background] Visser JE, Carpenter MG, van der Kooij H, Bloem BR. The clinical utility of posturography. Clin Neurophysiol. 2008 Nov;119(11):2424-36. doi: 10.1016/j.clinph.2008.07.220. Epub 2008 Sep 12. PMID 18789756
- [Background] Scaglioni-Solano P, Aragon-Vargas LF. Validity and reliability of the Nintendo Wii Balance Board to assess standing balance and sensory integration in highly functional older adults. Int J Rehabil Res. 2014 Jun;37(2):138-43. doi: 10.1097/MRR.0000000000000046. PMID 24445863
- [Background] Kwok BC, Clark RA, Pua YH. Novel use of the Wii Balance Board to prospectively predict falls in community-dwelling older adults. Clin Biomech (Bristol). 2015 Jun;30(5):481-4. doi: 10.1016/j.clinbiomech.2015.03.006. Epub 2015 Mar 11. PMID 25796535
- [Background] Johansson J, Nordstrom A, Nordstrom P. Objectively measured physical activity is associated with parameters of bone in 70-year-old men and women. Bone. 2015 Dec;81:72-79. doi: 10.1016/j.bone.2015.07.001. Epub 2015 Jul 4. PMID 26151120
- [Background] Johansson J, Nordstrom A, Nordstrom P. Greater Fall Risk in Elderly Women Than in Men Is Associated With Increased Gait Variability During Multitasking. J Am Med Dir Assoc. 2016 Jun 1;17(6):535-40. doi: 10.1016/j.jamda.2016.02.009. Epub 2016 Mar 19. PMID 27006336
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] Yardley L, Beyer N, Hauer K, Kempen G, Piot-Ziegler C, Todd C. Development and initial validation of the Falls Efficacy Scale-International (FES-I). Age Ageing. 2005 Nov;34(6):614-9. doi: 10.1093/ageing/afi196. PMID 16267188
- [Background] Tinetti ME, Richman D, Powell L. Falls efficacy as a measure of fear of falling. J Gerontol. 1990 Nov;45(6):P239-43. doi: 10.1093/geronj/45.6.p239. PMID 2229948
- [Derived] Sorlen N, Hult A, Nordstrom P, Nordstrom A, Johansson J. Short-term balance training and acute effects on postural sway in balance-deficient older adults: a randomized controlled trial. BMC Sports Sci Med Rehabil. 2021 Mar 9;13(1):23. doi: 10.1186/s13102-021-00251-x. PMID 33750421

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2017-07-13): https://cdn.clinicaltrials.gov/large-docs/66/NCT03227666/Prot_SAP_000.pdf
  • Informed Consent Form: Intervention (2017-05-11): https://cdn.clinicaltrials.gov/large-docs/66/NCT03227666/ICF_001.pdf
  • Informed Consent Form: Control (2017-05-11): https://cdn.clinicaltrials.gov/large-docs/66/NCT03227666/ICF_002.pdf